CLINICAL TRIAL: NCT06796062
Title: A Phase 2 Trial of Psilocybin as an Adjunctive Treatment for OUD Patients Who Continue to Use Illicit Opioids Despite Adherence to Methadone Treatment
Brief Title: Psilocybin for Opioid Use Disorder (OUD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-01120; 1UG3DA062088-01 (NIH)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Stage 1: Psilocybin 30 mg (high dose) (Experimental): Participants will receive a single IP administration (30 mg) session and remain under supervision at the facility for 8 hours.
  Interventions: Drug: Psilocybin
- Stage 1: Psilocybin 20 mg (medium dose) (Experimental): Participants will receive a single IP administration (20 mg) session and remain under supervision at the facility for 8 hours.
  Interventions: Drug: Psilocybin
- Psilocybin 1 mg (control) (Active Comparator): Participants will receive a single IP administration (1 mg) session and remain under supervision at the facility for 8 hours.
  Interventions: Drug: Psilocybin
- Stage 2: Psilocybin 30 mg (high dose) (Experimental): Participants will receive a single IP administration (30 mg) session and remain under supervision at the facility for 8 hours.
  Interventions: Drug: Psilocybin
- Stage 2: Psilocybin 20 mg (medium dose) (Experimental): Participants will receive a single IP administration (20 mg) session and remain under supervision at the facility for 8 hours.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — One capsule (1 mg, 20 mg, or 30 mg) administered once orally

SUMMARY:
This is a double-blind, adaptive, 2-stage, multi-site, phase 2 randomized controlled clinical trial designed to evaluate effects of moderate and high dose psilocybin, relative to low-dose psilocybin control, in OUD patients who continue to use illicit opioids in spite of adherence to standard-of-care treatment with methadone. Up to 480 participations will be consented to yield 240 randomized participants. This study is part of the NIH HEAL Initiative (https://heal.nih.gov/).

In Stage 1, subjects will be randomly assigned to one of three groups: psilocybin 30 mg (high dose), psilocybin 20 mg (medium dose), and psilocybin 1 mg (control condition). By the end of Stage 1, an interim statistical analysis will be performed. The study will proceed to Stage 2 if at least one of the active dosages of psilocybin demonstrates 1) acceptable safety, based on analysis of safety data from Stage 1; and 2) conditional power of at least 25%, based on effect size estimates for the primary opioid use outcome (weeks of biologically-verified abstinence during 24 weeks of follow-up). Using a priori decision rules, the interim analysis will determine which of the active treatment groups (30 mg, 20 mg, or both) will be retained in Stage 2 of the trial. Stage 2 will continue the study, using the same treatment and assessment protocols, but retaining only the active dosage or dosages with a high probability of demonstrating efficacy relative to the psilocybin 1 mg control condition.

The primary aims are to 1) Evaluate safety and efficacy outcomes in Stage 1 subjects in order to optimize design of the Stage 2, 2) Determine whether treatment with a single high (30 mg) or medium (20 mg) dose of psilocybin improves OUD treatment outcomes, relative to psilocybin 1 mg (control condition), in patients who continue to use illicit opioids despite adherence to methadone treatment, 3) Evaluate the effects of high-dose psilocybin and medium dose psilocybin on self-reported OUD-related neuropsychopathology, and 4) Identify likely responders to psilocybin treatment by using machine learning to model post-treatment OUD outcomes, based on pretreatment characteristics including all relevant clinical data, evaluations, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Are able to provide voluntary informed consent.
2. Have a breath alcohol concentration ≤ 0.01% at Screening Part 2, as determined by a breath alcohol reading from a calibrated breath alcohol sensor. (Note: this criterion may be re-evaluated within the 30-day screening period. This criterion will also be reassessed at Baseline and on Day 0 (prior to IP administration). Those not meeting the criterion may be rescheduled once within 14 days if the criterion is likely to resolve within 14 days in the judgement of the Investigator).
3. Are able to read, speak, and understand English, as documented during the informed consent process.

   a. Non-English speaking subjects will be excluded because the study is using only validated English-language versions of of assessment instruments.
4. Are 18 to 65 years old, inclusive, at Screening Part 2.
5. Have Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM 5) diagnosis of OUD, based on an evaluation performed by trained study staff using the Mini-International Neuropsychiatric Interview (MINI).
6. Want to stop their use of illicit opioids.
7. Are in treatment at one of participating Opioid Treatment Programs (OTPs) for at least 6 months at the time of Screening Part 2.
8. Are currently prescribed a methadone dose of at least 60 mg per day.
9. Methadone dosage has changed by no more than 20 mg in the past month
10. Have taken methadone at least 25 out of the last 30 days
11. Have had at least one urine drug screen positive for non-prescribed opioids in the past 30 days at the time of Screening Part 2
12. Report using opioids by insufflation, injection, or smoking
13. Are able and willing to adhere to all study requirements, including attending all study visits and treatment sessions, and completing all assessments.
14. Are able to provide at least one drug screen negative for illicit opioids, cocaine, and amphetamine-type stimulants during the screening period. (Note: this criterion may be re-evaluated within the 30-day screening period. This criterion will be reassessed at Day 0 [prior to IP administration]. Those not meeting the criterion on Day 0 may be rescheduled within 14 days if the criterion is likely to resolve in the judgement of the Investigator.)
15. Agree to refrain from any non-prescribed psychotropic substance or illicit drug use for at least 72 hours prior to IP administration, with the exceptions of alcohol, cannabis, nicotine, and caffeine. Regarding alcohol and cannabis, subjects must agree to attempt to abstain at least 24 hours before the IP administration session. Regarding nicotine, they must agree not to use nicotine for at least 1 hour before and 6 hours following IP administration. Regarding caffeine, they must agree to consume approximately their usual amount of caffeine on the morning of Day 0 (prior to IP administration).
16. Agree to refrain from taking all non-prescription medications and supplements (nutritional and herbal) for at least 1 week prior to the IP administration session unless approved by the Investigator.
17. Are able to swallow capsules.
18. Agree to practice effective contraception as described below.

    1. Subjects are considered able to become pregnant unless they:

       * Do not have a uterus
       * Are postmenopausal (has had 12 months of natural amenorrhea with a matching clinical profile [age, history of vasomotor symptoms]) prior to Screening Part 2, or
       * Are surgically sterile (documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy)
    2. Subjects who are able to become pregnant must:

       * Have a negative pregnancy test at Screening Part 2 (Reassessed at Day 0 (pre-IP administration);
       * Not be currently breastfeeding;
       * Not intend to become pregnant during participation in this study;
       * Agree to use a highly effective form of contraception from the time of the Screening Part 2 until 7 days after the IP Administration Session. Highly effective forms of contraception include: 1) Consistent and correct usage of established oral contraception; 2) Injected or implanted hormonal methods of contraception; 3) Established intrauterine device or intrauterine system; 4) Bilateral tubal ligation; 5) Intercourse with a partner who has undergone effective surgical sterilization, provided that partner is the sole sexual partner of the study subject; 6) Abstinence from penile/vaginal intercourse, if the Investigator determines that the subject can reliably adhere to the plan, based on evaluation of the social circumstances of the subject.
    3. Agree not to donate or bank eggs from the time of Screening Part 2 until 7 days after the IP Administration Session.
    4. Subjects who can emit sperm are defined as those who:

       * Have one or more testes and
       * Have not had a documented effective surgical sterilization procedure (e.g., vasectomy, radical prostatectomy).
    5. Subjects who can emit sperm must:

       * Practice effective contraception from Screening Part 2 until 7 days after the IP Administration Session. Effective means forms of contraception include:
       * use condoms with spermicide if engaging in penile/vaginal intercourse;
       * abstain from penile/vaginal intercourse, if the Investigator determines that the subject can reliably adhere to the plan, based on evaluation of the social circumstances of the subject
       * Agree not to donate or bank sperm from the time of the Screening Part 2 until 7 days after the IP Administration Session
19. Have a family member or friend who can assist with transportation and activities of daily living after the IP Administration Session, as determined by self-report at Screening Part 2 and confirmed by direct communication between a member of the clinical support team and the support person prior to randomization. (Note: this criterion will be reassessed on Day 0.
20. Are able to provide adequate locator information. This criterion may be re-evaluated within the 30-day screening period.

Exclusion Criteria:

1. Have any medical condition that would preclude safe participation in the study, including the following, as determined by medical history review, physical examination, electrocardiogram (ECG), and clinical laboratory tests:

   1. Seizure disorder
   2. Significantly impaired liver function, defined as 1) alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 5 × upper limit of normal (ULN); 2) ALT or AST > 3 × ULN with concomitant total bilirubin > 2.0 × ULN; or 3) ALT or AST ≥ 3 × ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia.
   3. Cardiovascular disease including coronary artery disease, angina, history of arrhythmia (unless a successful ablation has been performed), heart failure, history of heart valve replacement, and history of cerebrovascular accident or transient ischemic attack.
   4. Uncontrolled hypertension with systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg. (Note: subjects who otherwise qualify at Screening Part 2 will have 3 opportunities to produce 1 blood pressure reading ≤ 140/90 mmHg (each reading will be collected at least 15 minutes apart). If blood pressure is consistently elevated > 140/90 mmHg across all 3 attempts, subjects may be referred to their primary care provider for management of hypertension. Upon management of blood pressure, subjects will have an opportunity to return once within the 30 day screening window to make 3 additional attempts at a blood pressure reading ≤ 140/90 mmHg. Subjects will be considered eligible upon registering 1 blood pressure reading ≤ 140/90 mmHg during the screening period. Blood pressure will be reassessed on Day 0 prior to dosing, and must be less than or equal to 140 systolic, 90 diastolic, with resting pulse ≤ 100 (ascertained within 20 minutes of drug administration in order for the participant to receive study medication.)
   5. Serious ECG abnormalities present on the ECG obtained on Day -65 (e.g., evidence of ischemia, myocardial infarction, QT interval corrected for heart rate [QTc] prolongation (QTc > 0.45 seconds), arrhythmia, or conduction abnormalities that increase the risk of arrhythmia.
   6. Hyperthyroidism
   7. Insulin-dependent diabetes
   8. Any other medical condition which precludes safe participation in the study in the medical opinion of the Investigator.

   (Note: medical history will be updated and ECG will be repeated on Day 0, prior to dosing. Those not meeting the criterion will not be randomized but may be rescheduled once within 14 days if the criterion is likely to resolve within 14 days in the judgement of the Investigator.)
2. Have any of the following DSM-5 psychiatric disorders, as determined by the MINI, Psychiatric History and Psychosis Screening Questionnaire at Screening Part 2: (Note: psychiatric history will be re-evaluated on Day 0, but the MINI will not be re-administered on Day 0)

   1. Lifetime history of schizophrenia spectrum or other psychotic disorder.
   2. Lifetime history of bipolar disorder.
   3. Current severe major depression (based on a MINI diagnosis of major depression, current, and a MADRS score >34 at Screening)
   4. Alcohol use disorder including alcohol withdrawal.
   5. More than mild opioid withdrawal (COWS score >12). (This criterion may be re-evaluated within the 30-day screening period. This criterion will be reassessed on Day 0. Those not meeting the criterion may be rescheduled once within 14 days if the criterion is likely to resolve within 14 days in the judgement of the Investigator.)
3. Have active suicidal ideation with intent, based on Columbia - Suicide Severity Rating Scale (C-SSRS) assessment (severity score >3) at Screening Part 2, confirmed by the Investigator. (Note: this criterion will be reassessed at each visit that occurs prior to Day 0, and on Day 0 prior to IP administration. Subjects will be discharged if actively suicidal, and appropriate follow-up will be arranged.arranged.
4. Have made a suicide attempt within the past 12 months, based on C-SSRS assessment at Screening Part 2 and confirmation by the Investigator. (Note: this criterion will be reassessed at each visit that occurs prior to Day 0, and on Day 0 prior to IP administration. Subjects will be discharged if actively suicidal, and appropriate follow-up will be arranged.
5. Have a family history (first degree relatives) of schizophrenia, schizoaffective disorder, or bipolar disorder type 1.
6. Have a history of hallucinogen use disorder or hallucinogen persisting perception disorder (HPPD).
7. Have any hallucinogen use in the past 1 year.
8. Have > 25 lifetime uses of classic psychedelics.
9. Are currently in jail, prison, or other overnight facility as required by court of law or have pending legal action that could prevent participation in study activities.
10. Are taking any protocol-prohibited medications and supplements (See Section 6.5.3). Any prohibited medications and supplements must have been stopped for at least 5 elimination half-lives or 14 days, whichever is longer, prior to Day 0. Prescribed psychotropic medications and any other medically necessary medications must not be stopped in order to qualify for the study. (Note: concomitant medications will be reassessed on Day 0.)
11. Have a known allergy or hypersensitivity to psilocybin or any of the materials contained in the IP used in the study.
12. Have an allergy, hypersensitivity, or other contraindication that would preclude safe treatment of acute hypertension, anxiety, or psychotic symptoms if necessary during or immediately after the IP Administration Session, using the adjunctive medications used in this study to treat these symptoms (i.e., unable to take captopril and unable to take clonidine; unable to take diazepam and unable to take lorazepam; or unable to take olanzapine).
13. Have any other medical, psychiatric, or psychosocial disorder, symptom, condition, or situation that is likely to interfere with the establishment of rapport, adherence to study requirements, or safe administration of psilocybin, based on the judgement of the Investigator. (Note: This criterion will be reassessed on Day 0. Those not meeting the criterion will not be randomized but may be rescheduled once within 14 days if the criterion is likely to resolve within 14 days in the judgement of the Investigator.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Stage 1: The number of weeks during the 24 week follow-up period with no illicit opioid use | Up to 24 weeks
  Subject reports no illicit opioid use and provides a urine drug screen (UDS) negative for all classes of opioids other than methadone or other legally prescribed opioids.
Stage 1: Number of adverse events | Up to 24 weeks
Stage 1: Change in QTc during drug administration session | Up to 24 weeks
Stage 2: The number of weeks during the 24 week follow-up period with no illicit opioid use | Up to 24 weeks
Stage 2: Number of adverse events | Up to 24 weeks
Stage 2: Change in QTc during drug administration session | Up to 24 weeks
Stage 2: Total score on the Penn Craving Scale for Opioids | Up to 24 weeks
  The Penn Alcohol Craving Scale (PACS) is a 5-item questionnaire that measures an individual's craving to drink alcohol in the past week. The self-report measure includes questions about the frequency, intensity, and duration of craving, the ability to resist drinking, and asks for an overall rating of craving for alcohol for the previous week. Each question is scaled from 0 to 6. Low score (below 15) indicates minimal to no reported alcohol craving. Moderate score (15-20) suggests a moderate level of alcohol craving. High score (above 20) represents a high level of alcohol craving, potentially warranting further assessment and treatment
Stage 2: Score on the Negative Affect subscale of the Positive and Negative Affect Scale | Up to 24 weeks
  The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point verbal frequency scale of 1 (not at all) to 5 (very much). Scores range from 10 - 50 for both sets of items. For the total negative score, a lower score indicates less of a negative affect.
Stage 2: Total score on the 20-item version of the Short Urgency, Premeditation, Perseverance, Sensation seeking, and Positive urgency (UPPS-P) Impulsive Behavior Scale (SUPPS-P) | Up to 24 weeks
  The 20-item version of the UPPS-P Impulsive Behavior Scale, also known as the SUPPS-P, is a shortened questionnaire that assesses five different dimensions of impulsivity: negative urgency, positive urgency, lack of perseverance, lack of premeditation, and sensation seeking; with four items dedicated to each dimension, totaling 20 questions in total. Responses are rated on a Likert scale (e.g., strongly disagree to strongly agree), with higher scores generally indicating a greater tendency towards impulsive behavior.

SECONDARY OUTCOMES:
Stage 2: Time to opioid relapse | Up to 24 weeks
  Defined as the number of days from the day of investigational product (IP) administration to a day of opioid use which marked the start of a) 4 consecutive opioid use weeks or b) the start of 7 consecutive days of self-reported opioid use days (ranging from 0 to 168 days).
Stage 2: Time to first illicit opioid use | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bogenschutz, MD, Principal Investigator — NYU Langone Health
Locations (5):
- United States (5):
  - Duke City Recovery Toolbox, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - StartCare, Brooklyn, New York
  - NYU Langone Health, New York, New York
  - VIP Community Services, Inc, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request immediately following publication, no end date, provided the investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. The NDA provides basic descriptive and aggregate summary information for general public use. Such summary information may include summary counts and general statistics on completed assessment instruments. Access to subject level datasets submitted and stored in the NDA will only be provided for research purposes through the completion of the NDA Data Use Certification: OMB Control Number: 0925-0667. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Access to subject level datasets submitted and stored in the The National Institute of Mental Health (NIMH) Data Archive (NDA) will only be provided for research purposes through the completion of the NDA Data Use Certification: Office of Management and Budget (OMB) Control Number: 0925-0667. For the majority of the data available in the NDA, Data Use Certifications will only be accepted from researchers who are sponsored by an institution registered in the NIH's Electronic Research Administration (eRA) Commons with an active Federal-wide Assurance issued through the Office for Human Research Protections (OHRP). Additionally, the application must include a reason for access related to scientific investigation, scholarship or teaching, or other form of research. A Data Access Committee (DAC) composed of NIH staff with relevant expertise reviews the Data Use Certification and makes decisions about whether to grant access to subject level data.